CLINICAL TRIAL: NCT02528760
Title: To Determine the Role of Prokinetics in Feed Intolerance in Critically Ill Cirrhosis- A Randomized Placebo Controlled Study
Brief Title: To Determine the Role of Prokinetics in Feed Intolerance in Critically Ill Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-005
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2016-09

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Metoclopramide; Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metaclopromide group (Experimental)
  Interventions: Drug: Metaclopramide
- Erythromycin group (Experimental)
  Interventions: Drug: Erythromycin
- Placebo group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metaclopramide — 23. Metoclopromide to be given 10mg iv 8 hourly
  Arms: Metaclopromide group
Drug: Erythromycin — Erythromycin to be given 70mg iv 12 hourly.
  Arms: Erythromycin group
Other: Placebo
  Arms: Placebo group

SUMMARY:
1. All patients with chronic liver disease admitted in ICU (Intensive Care Unit) to be screened.
2. Patients fulfilling criteria for feed intolerance to be included in the study.
3. Patients to undergo routine biochemical and hematological testing including CBC, KFT, LFT, PT/INR, electrolytes baseline and daily along with ABG (Arterial Blood gas) analysis.
4. Patients with ascites to be tested for presence or absence of SBP (Spontaneous Bacterial Peritonitis).
5. Cultures to be sent as based on clinical parameter of the patient.
6. All correctable causes for intra abdominal hypertension to be corrected including electrolyte imbalance, grade III ascites, intra abdominal infection.
7. Symptoms- Absent bowel sounds (BS)= no BS detected by auscultation. Vomiting/regurgitation= any visible regurgitation of gastric contents; Diarrhoea= liquid stool > or =3 times/day; Bowel distension= suspected clinically and radiologically confirmed; Large gastric residual volume (GRV) of >or =500 ml/24 h on a single day or > 200ml at any time of the day.
8. Per abdomen findings to be checked daily including presence of bowel sounds, tenderness, development of abdominal distension, abdominal girth monitoring and abdominal pressure monitoring.
9. Patients who develop feed intolerance will be included.
10. Feed intolerance to be defined as per study definition (3 out of 5 symptoms).
11. Measurement of GRV (Gastric residual volume) to be done at 4 hourly interval.
12. Methods for measuring GRV by either gravity drainage by connecting a gastric tube to a drainage bag for 10min or by manual aspiration of content using a 50ml syringe.
13. Once feed intolerance develop than every 6 hourly intra abdominal pressure monitoring and abdominal girth monitoring to be done (24)
14. Intra bladder pressure to be measured using Foleys manometer technique (25).
15. Pressure measured in cm of water to be converted into mm of Hg.
16. X ray abdomen supine to look for bowel distension, defined as more than 3 cm for small bowel and more than 5 cm in large bowel.
17. Development of intra abdominal hypertension based on intra abdominal pressure.
18. Patient to be stratified according to the grade of intra-abdominal hypertension.
19. After correction of all correctable causes, if feed intolerance persists, then patient to be randomized by block randomization method into 3 arms, metaclopromide group, erythromycin group or placebo group.
20. Daily assessment of bowel sounds, abdominal pressure, abdominal girth every 6 hourly and gastric residual volume to be noted every 4 hourly.
21. Response of therapy to be assessed at 24 hours in each arm.
22. Response to be assessed by resolution of feed intolerance or initiation of entral nutrition.
23. Metoclopromide to be given 10mg iv 8 hourly.
24. Erythromycin to be given 70mg iv 12 hourly (26).
25. Placebo arm to receive normal saline in 10ml syring twice daily.
26. After 24 hours of treatment if symptoms do not resolve than rescue treatment will be given to each arm which may include continuation of prokinetics, add on prokinetic, flatus tube insertion for bowel decompression, upgradation of antibiotics or search for any other cause, as per the patient response.
27. Therapy to continue for a total duration of 72 hours.
28. If there is no response at 72 hours, than study stops.
29. If patient responds to given treatment, study to continue for a total duration of 7 days.
30. Assessment to continue in each arm for a maximum period of 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who develop new onset feed intolerance to enteral nutrition

Exclusion Criteria:

1. Any patient with current or past surgical abdomen including mechanical obstruction, mesenteric ischemia, perforation or requiring abdominal surgery.
2. Patients receiving enteral nutrition through gastrostomy or jejunostomy.
3. Patients in whom, prokinetics are contraindicated or are allergic to the same.
4. Patients who received prokinetic more than one day prior to the start of enteral feeding.
5. Patients with uncontrolled sepsis with DIC.
6. Requirement of two or more vasopressors.
7. Organ failure requiring high inotropic support.
8. Advanced cardiopulmonary disease, with prior history of arrhythmias, structural heart disease.
9. History of traumatic brain injury, raised intracranial pressure, history of myasthenia gravis.
10. Endocronolgic illnesses: Hypothyroidism, hypoparathyroidism
11. Connective tissue diseases (systemic sclerosis, dermatomyositis or polymyositis, systemic lupus erythematosis, amyloidosis).
12. Known case of diabetes with diabetic gastroparesis
13. Pregnancy
14. Patients or concerned family member who fail to give consent for study enrollment
15. Age less than 18 years and more than 70 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Resolution of feed intolerance at 24 hours with improvement in 3 or more points and initiation of entral feeding. | 24 hours
  Feed intolerance to be defined as 3/5 symptoms which include gastric residual volume > 500 ml /day,absence of bowel sounds,vomitting/regurgitation,diarrhoea and bowel distension

SECONDARY OUTCOMES:
Survival | 72 hours
Survival | 7 days
Number of patients with Initiation of entral nutrition more than 50%. of recommended nutrition (Kcal/kg body weight/day). | 72 hours
  Feed intolerance is also defined when entral nutrition provided < 20Kcal/kg body weight/day.
Number of patients with resolution of atleast 2 out of 5 symptoms in all the 3 groups. | 72 hours
  Feed intolerance to be defined as 3/5 symptoms which include gastric residual volume > 500 ml /day,absence of bowel sounds,vomitting/regurgitation,diarrhoea and bowel distension
Number of patients with resolution of sepsis, shock, organ failure in all the 3 groups. | 7 days
Number of patients without Ventilatory support in all the 3 groups. | 7 days
Number of patients without inotropic supports in all the 3 groups. | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India